CLINICAL TRIAL: NCT04832854
Title: A Phase II, Open-Label, Multicenter Study Evaluating the Safety and Efficacy of Neoadjuvant and Adjuvant Tiragolumab Plus Atezolizumab, With or Without Platinum-Based Chemotherapy, in Patients With Previously Untreated Locally Advanced Resectable Stage II, IIIA, or Select IIIB Non-Small Cell Lung Cancer
Brief Title: A Study Evaluating the Safety and Efficacy of Neoadjuvant and Adjuvant Tiragolumab Plus Atezolizumab, With or Without Platinum-Based Chemotherapy, in Participants With Previously Untreated Locally Advanced Resectable Stage II, IIIA, or Select IIIB Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO42501; 2020-002853-11 (EudraCT Number)
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Tiragolumab; Carboplatin; Cisplatin; Pemetrexed; Gemcitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (PD-L1 High) (Experimental): Participants with high programmed death-ligand 1 (PD-L1) expression level will be enrolled in Cohort A and receive neoadjuvant atezolizumab plus tiragolumab for 4 cycles, followed by surgical resection and either adjuvant atezolizumab plus tiragolumab for 16 cycles or adjuvant chemotherapy for 4 cycles at the discretion of the investigator.
  Chemotherapy may include:
  * cisplatin/carboplatin + pemetrexed (for non-squamous only)
  * carboplatin + gemcitabine (for squamous only)
  * carboplatin + paclitaxel
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed; Drug: Gemcitabine; Drug: Paclitaxel
- Cohort B (PD-L1 All Comers) (Experimental): All comers, which are participants with any PD-L1 expression level, will be enrolled in Cohort B and receive neoadjuvant atezolizumab plus tiragolumab plus chemotherapy for 4 cycles, followed by surgical resection and adjuvant atezolizumab plus tiragolumab for 16 cycles.
  Chemotherapy may include:
  * cisplatin/carboplatin + pemetrexed (for non-squamous only)
  * carboplatin + gemcitabine (for squamous only)
  * carboplatin + paclitaxel
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed; Drug: Gemcitabine; Drug: Paclitaxel

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg will be administered by intravenous (IV) infusion on Day 1 of each 21-day cycle.
  Other Names: Tecentriq
Drug: Tiragolumab — Tiragolumab 600 mg will be administered by IV infusion on Day 1 of each 21-day cycle.
  Other Names: MTIG7192A
Drug: Carboplatin — Carboplatin at initial target area under the concentration curve (AUC) of 5 or 6 mg/mL/min will be administered by IV infusion on Day 1 of each 21-day cycle.
Drug: Cisplatin — Cisplatin at 75 mg/m^2 will be administered by IV infusion on Day 1 of each 21-day cycle.
Drug: Pemetrexed — Pemetrexed at 500 mg/m^2 will be administered by IV infusion on Day 1 of each 21-day cycle.
Drug: Gemcitabine — Gemcitabine at 1000 or 1250 mg/m^2 will be administered by IV infusion on Days 1 and 8 of each 21-day cycle.
Drug: Paclitaxel — Paclitaxel at 175 or 200 mg/m^2 will be administered by IV infusion on Day 1 of each 21-day cycle.

SUMMARY:
This study will evaluate the surgical safety and feasibility of atezolizumab plus tiragolumab alone or in combination with platinum-based chemotherapy as neoadjuvant treatment for participants with previously untreated locally advanced non-small cell lung cancer (NSCLC). The study will also evaluate the efficacy, pharmacokinetics, immunogenicity, and safety of atezolizumab plus tiragolumab alone or in combination with platinum-based chemotherapy as neoadjuvant treatment, followed by adjuvant atezolizumab plus tiragolumab or adjuvant platinum-based chemotherapy.

ELIGIBILITY:
Key inclusion criteria:

* Histologically or cytologically confirmed Stage II, IIIA, or select IIIB (T3N2 only) NSCLC of squamous or non-squamous histology
* Eligible for R0 resection with curative intent at the time of screening
* Adequate pulmonary function to be eligible for surgical resection with curative intent
* Eligible to receive a platinum-based chemotherapy regimen
* Measurable disease, as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Availability of a representative tumor specimen that is suitable for determination of PD-L1 status
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Normal life expectancy, excluding lung cancer mortality risk
* Adequate hematologic and end-organ function
* Negative human immunodeficiency virus (HIV) test at screening
* Negative serology for active hepatitis B virus (HBV) and active hepatitis C virus (HCV) at screening

Key Exclusion Criteria:

* NSCLC with histology of large cell neuroendocrine carcinoma, sarcomatoid carcinoma, or NSCLC not otherwise specified
* Small cell lung cancer (SCLC) histology or NSCLC with any component of SCLC
* Any prior therapy for lung cancer
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Active tuberculosis
* Significant cardiovascular disease
* NSCLC with an activating EGFR mutation or ALK fusion oncogene
* Known c-ros oncogene 1 (ROS1) rearrangement
* History of malignancy other than NSCLC within 5 years prior to screening, with the exception of malignancies with negligible risk of metastasis or death
* Severe infection within 4 weeks prior to initiation of study treatment or any active infection that, in the opinion of the investigator, could impact patient safety
* Prior treatment with CD127 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, anti-TIGIT, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents
* Treatment with systemic immunosuppressive medication
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Surgical Delays | Up to approximately 6 years
Number of Participants With Operative and Post-operative Complications | Up to approximately 6 years
Number of Participants With Surgical Cancellations Related to Study Treatment | Up to approximately 6 years
Percentage of Participants With Adverse Events | Up to approximately 6 years
Percentage of Participants Who Achieve Major Pathological Response (MPR) | At the time of surgery (approximately Weeks 17-20)

SECONDARY OUTCOMES:
Percentage of Participants With Pathological Complete Response (pCR) | At the time of surgery (approximately Weeks 17-20)
Event Free Survival (EFS) | From baseline to disease progression that precludes surgical resection, or local or distant disease recurrence after surgery, or death from any cause (up to approximately 6 years)
Serum Concentrations of Atezolizumab | Day 1 of Cycle 1 (cycle=21 days): pre-dose and 30 minutes (min) post-dose; Day 1 of Cycles 2, 3, 4, 5, 8, 12, 16: pre-dose; at treatment discontinuation (TD) visit (up to approximately 9 months)
Serum Concentrations of Tiragolumab | Day 1 of Cycle 1 (cycle=21 days): pre-dose and 30 min post-dose; Day 1 of Cycles 2, 3, 4, 5, 8, 12, 16: pre-dose; at TD visit (up to approximately 9 months)
Percentage of Participants With Anti-drug Antibodies (ADAs) to Atezolizumab | Prior to the first infusion on Day 1 of Cycles 1, 2, 3, 4, 5, 8, 12 and 16 (cycle=21 days) and at TD visit (up to approximately 9 months)
Percentage of Participants With ADAs to Tiragolumab | Prior to the first infusion on Day 1 of Cycles 1, 2, 3, 4, 5, 8, 12 and 16 (cycle=21 days) and at TD visit (up to approximately 9 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- United States (7):
  - City of Hope Cancer Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - University of Southern California, Los Angeles, California
  - Washington University School of Medicine, St Louis, Missouri
  - Winthrop Univ Hospital, Mineola, New York
  - NYU Cancer Center, New York, New York
  - Columbia University, New York, New York
- Australia (2):
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Peter Maccallum Cancer Institute, Melbourne, Victoria
- South Korea (2):
  - St. Vincent's Hospital, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (6):
  - ICO L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- Switzerland (5):
  - Kantonsspital Baden, Baden
  - Kantonsspital Graubünden Medizin Onkologie, Chur
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - UniversitätsSpital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing